CLINICAL TRIAL: NCT02244905
Title: Trial of Positive Deviance in Inpatient Wards to Reduce Hospital Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU 072011-079; Grant # 137911 (Other: University of Texas System Patient Safety)
Record Dates: First submitted 2014-09-15; First posted 2014-09-19 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Healthcare-associated Infections
Keywords: Positive Deviance; Infection Control; Healthcare-Associated Infections; Staff Engagement; Cluster Randomized Controlled Trial
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Positive Deviance Intervention Arm (Experimental): Three hospital wards received Positive Deviance intervention.
  Interventions: Behavioral: Positive Deviance; Other: Standard-of-Care Infection Control approach
- Control Arm (Other): Three hospital wards randomized to control arm received the Standard-of-Care Infection Control approach.
  Interventions: Other: Standard-of-Care Infection Control approach

INTERVENTIONS:
Behavioral: Positive Deviance — The recipients of the Positive Deviance intervention are the staff members of the three wards in the intervention arm, while the outcomes are measured among the patients receiving care in the three wards in the intervention arm. Key components of the intervention were invitation to participate voluntarily, open-ended dialogues with staff members to discover barriers and seek solutions to prevent HAI, discussion of outcomes, and encouragement to prioritize and implement the solutions generated.
  Arms: Positive Deviance Intervention Arm
Other: Standard-of-Care Infection Control approach — Standard-of-Care Infection Control approach

SUMMARY:
Healthcare-associated infections (HAI) are a significant public health burden. Even with existence of recommendations on technical strategies to prevent these infections, there is a need for strategies to increase staff engagement within the local organizational and cultural context. Positive deviance is one such approach that engages people in improvement efforts. Positive Deviance is based on the observation that in every community there are certain individuals or groups whose uncommon behaviors and strategies enable them to find better solutions to problems than their peers, while having access to the same resources and facing similar or worse challenges. In the proposed study, the investigators plan to test the effectiveness of using positive deviance based horizontal infection prevention approach to achieve overall reduction of HAIs among hospital inpatients. The investigators hypothesized that a broad and horizontal approach to reduce opportunities for acquisition of nosocomial pathogens using PD will lead to greater reduction of HAI among hospital inpatients compared to standard-of-care infection control approach. The investigators objective was to test the investigators hypothesis and evaluate whether there is greater decline in rate of HAI in the experimental group of wards compared to the control group of wards.

DETAILED DESCRIPTION:
Objective: To evaluate whether positive deviance (PD) based horizontal infection prevention approach will result in a higher rate of decline in incidence density of patients with HAI (central line-associated bloodstream infection, healthcare-associated pneumonia, catheter-associated urinary tract infection, or Clostridium difficile infection) per 1000 patient days per month in the intervention wards compared to control wards.

Design: A cluster randomized controlled trial was conducted over a period of 24 months. Six medical wards were randomized and positive deviance intervention was randomly allocated to one of the two groups of three wards each. The baseline, intervention and follow-up periods were 6, 9 and 9 months respectively.

Setting: A public safety-net major teaching hospital in United States.

Participants: The ward staffs participated in the intervention.

Intervention: Key components of the intervention were invitation to participate voluntarily, open-ended dialogues with staff members to discover barriers and seek solutions to prevent HAI, discussion of outcomes, and encouragement to prioritize and implement the solutions generated. Staffs of all six wards were asked to voluntarily participate in a modified hospital survey of patient safety climate (HSOPSC) and a social network survey at 6, 15, and 24 months.

Statistical analysis: Statistical methods used were time series modeling, summary of frequencies, Chi-square or Fisher's exact for testing difference in proportions and t-test.

ELIGIBILITY:
The intervention was performed on the staff members providing care in the three wards belonging to the intervention arm of the study. These staff members were invited to participate in the positive deviance intervention on a voluntary and anonymous basis.

The primary outcome was measured in all the patients who received care in the three intervention wards and the three control wards.

Inclusion Criteria:

* For Intervention: All staff members employed in the study wards assigned to the intervention arm.
* For Primary Outcome Assessment:

  * All patients admitted to any of the six study wards included in the study over the 24-month study period.

Exclusion Criteria:

-None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16876 (Actual)
Dates: Start 2011-08; Primary Completion 2013-03 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number of HAI per 1000 patient-days per month. | 24 Months
  The primary study outcome is the incidence density of HAI [a composite of central line associated bloodstream infection (CLABSI), hospital-acquired pneumonia (HAP), catheter-associated urinary tract infection (CAUTI) and C.difficile infection (CDI)] per 1000 patient-days per month.

CONTACTS AND LOCATIONS:
Overall Officials: Pranavi Sreeramoju, MD, Principal Investigator — University of Texas Southwestern Medical Center